CLINICAL TRIAL: NCT05069337
Title: Biobank of Lung Ultrasonography in Children Undergoing General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-1035
Record Dates: First submitted 2021-09-23; First posted 2021-10-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Children Aged 6 Months to 10 Years Old Under General Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For children aged 6 months to 10 years old under general anesthesia, intraoperative lung ultrasound pictures are acquired, grades are evaluated for each pictures and machine learning is used to learn and apply it.

DETAILED DESCRIPTION:
1. routine general anesthesia is performed in the selected children.
2. After mechanical ventilation, the degree of lung atelectasis is evaluated using transthoracic lung ultrasonography in the anterior, lateral, posterior regions of the upper and lower points of both lungs(a total of 12 regions).
3. Atelectasis is checked by the presence of B-line and juxta pleural consolidation.
4. Machine learning is used to educate the photos of 70 people and grading system, and process is checked whether it applies well to the photos of the remaining 30 people.

ELIGIBILITY:
Inclusion Criteria:

1. children aged 6 months to 10 years old under general anesthesia
2. ASA I-III

Exclusion Criteria:

1. If the parents of the patient cannot communicate in Korean
2. If mechanical ventilation is not planned (for example, A1 pulley)
3. emergency operation
4. a child whose ultrasound image quality is expected to deteriorate due to diseases such as thoracic deformity, scoliosis, or rib fractures
5. If lateral position was not available

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children aged 6 months to 10 years old under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
consolidation score | After intubation and before the surgery start or after the surgery complete and before the extubation
  Sum of the consolidation scores at 12 lesions by the lung ultrasonography

SECONDARY OUTCOMES:
B-line score | After intubation and before the surgery start or after the surgery complete and before the extubation
  Sum of the B-line scores at 12 lesions by the lung ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jin Byon, Principal Investigator — Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No